CLINICAL TRIAL: NCT03545334
Title: A Diagnostic Sensitivity Study Comparing Intradermal ICG and NIRFI With Intradermal Technetium 99m and Traditional Lymphoscintigraphy for Transcutaneous Identification of Sentinel Lymph Nodes in Malignant Melanoma
Brief Title: Lymph Node Identification in Skin Malignancy Using ICG Transcutaneously Study
Acronym: LIMIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KEK-Nr. 2016-01746
Record Dates: First submitted 2018-05-22; First posted 2018-06-04 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Malignant Melanoma; Merkel Cell Carcinoma
Keywords: transcutaneous identification of SLNs with ICG
MeSH Terms: conditions — Melanoma; Carcinoma, Merkel Cell

STUDY DESIGN:
Intervention Model Description: A diagnostic sensitivity study comparing intradermal indocyanine green (ICG) and near infrared fluorescence imaging (NIRFI) with intradermal technetium 99m and traditional lymphoscintigraphy (LS) for transcutaneous identification of sentinel lymph nodes (SLN) in malignant melanoma - a prospective Phase II clinical study in a single center.
Masking Description: The surgeons performing SLNB will be the blinded persons. The results of the lymphoscintigraphy will not be marked on the patient's skin as usual and no preoperative access to the images will be granted to the surgeons.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Comparison result lymphoscintigraphy with ICG lymphography (Experimental): The patient first receives a standard Tc-99m-based lymphoscintigraphy. The identified lymph nodes are not marked in the patients, so that the surgeons are not affected in lymph node identification during ICG and near infrared fluorescence imaging. The surgeon also has no access to lymphoscintigraphy images.
  Transcutaneous ICG lymphography is then performed by intradermal injection of ICG around the scar of the primary tumor excision and transcutaneous fluorescence evaluation with the Visionsense™ VS3 - Stereoscopic High Definition Visualisation System (VS3-3DHD) and results are compared.
  Interventions: Diagnostic Test: Visionsense™ VS3 - Stereoscopic High Definition Visualisation System (VS3-3DHD)

INTERVENTIONS:
Diagnostic Test: Visionsense™ VS3 - Stereoscopic High Definition Visualisation System (VS3-3DHD) — Injection of ICG intradermally around the scar of the primary excision of the tumour and transcutaneous assessment of fluorescence with the VS3-3DHD camera (Visionsense™ VS3 - Stereoscopic High Definition Visualisation System ).
  Other Names: Indocyanin green (ICG)

SUMMARY:
A diagnostic sensitivity study comparing intradermal indocyanine green (ICG) and near infrared fluorescence imaging (NIRFI) with intradermal technetium 99m and traditional lymphoscintigraphy (LS) for transcutaneous identification of sentinel lymph nodes (SLN) in malignant melanoma - a prospective Phase II clinical study in a single center.

DETAILED DESCRIPTION:
Switzerland has the highest rate of new melanomas in Europe (19.2 per 100,000). Melanomas have the worst prognosis of all skin cancers. The current treatment depends on the histological diagnosis after a biopsy and is primarily related to the tumor thickness (Breslow Score), the tumor cells in division (mitosis rate), the substance defect of the skin (ulceration), the occurrence of regression, and the age of the patients. The initial treatment is performed by surgical removal with a safety margin of macroscopically healthy skin around the tumor. If the tumor thickness is more than 1 mm or more than 0.7 mm associated with a high mitosis rate in younger patients, ulcerations, regression or Clark Level IV / V, then current melanoma guidelines suggest that the patient undergoes sentinel lymph node biopsy (SLKB) as this is most likely the first site where metastases spread. Merkel cell carcinoma is a very aggressive, neuroendocrine skin tumor with a mortality rate of about 33% after 3 years. Due to the frequent lymphatic metastases, SLNB is highly recommended in all patients in order to better assess their prognosis. The gold standard technique to identify SLKs is to inject the radioisotope Technetium-99m around the primary tumor into the skin. The patient is then scanned to determine the position of the SLK after approximately 30 and 120 minutes. Other teams have attempted to identify transcutaneous SLK with ICG and NIRFI, but have concluded that ICG fluorescence technique is not reliable in patients with high BMI or a primary tumor with lymph drainage in the axillary lymph node region. This study aims to evaluate a medical device that uses an improved technology compared to previous studies (stereoscopic 3D high definition for both fluorescence and visible light imaging). The investigators hope is that by applying similar principles SLKs can be identified through the use of transcutaneous fluorescent dye injections and NIRFI.

ELIGIBILITY:
Inclusion Criteria:

* Malignant melanoma patients having one of the following characteristics:

  * Breslow score ≥ 1 mm
  * Breslow score ≥ 0.7 mm associated with ulceration
  * Breslow score ≥ 0.7 mm associated with regression
  * Breslow score ≥ 0.7 mm associated with Clark Level IV / V
  * Breslow score ≥ 0.7 mm associated with mitotic rate ≥ 1/mm2 in young patients
* Merkel cell carcinoma

Exclusion Criteria:

* Age < 18 years
* Pregnancy and breastfeeding (pregnancy test to be performed for women of child-bearing potential, defined as women who are not surgically sterilized/ hysterectomized, and/or who are postmenopausal for less than 12 months)
* Known allergy to ICG or Iodine
* Previous chemotherapy, radiotherapy or surgery to the lymph nodes of interest
* Lack of capacity to provide informed consent
* Current enrolment in any other interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Correlation of sentinel lymph nodes identified by lymphoscintigraphy vs. VisionSense near-infrared-fluorescence-imaging. | one hour
  To determine whether the VisionSense NIRFI technology can transcutaneously identify SLNs as effectively as LS.

SECONDARY OUTCOMES:
Correlation of sentinel lymph nodes identified by lymphoscintigraphy vs. VisionSense near-infrared-fluorescence-imaging in specific anatomical locations and in defined patient groups (e.g. groups defined based on BMI, sex, age). | one hour
  The study seeks primarily to determine ability of the VisionSense NIRFI technology to transcutaneously identify SLNs as effectively as LS.

CONTACTS AND LOCATIONS:
Overall Officials: Mihai A. Constantinescu, Professor, Study Director — Clinic for Plastic and Reconstructive Surgery, Inselspital Bern, Switzerland; Radu Olariu, MD, Principal Investigator — Clinic for Plastic and Reconstructive Surgery, Inselspital Bern, Switzerland
Locations (1):
- Inselspital, University Hospital Bern, University of Bern, Bern, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lese I, Leckenby JI, Taddeo A, Constantinescu M, Olariu R. Lymph node identification in skin malignancy using indocyanine green transcutaneously study: Study protocol for a diagnostic accuracy study. Medicine (Baltimore). 2019 Nov;98(44):e17839. doi: 10.1097/MD.0000000000017839. PMID 31689874